CLINICAL TRIAL: NCT04514341
Title: Implementing a Multilevel Intervention to Accelerate Colorectal Cancer Screening and Follow-up in Federally Qualified Health Centers Using a Stepped Wedge Design
Brief Title: Implementing a Multilevel Intervention to Accelerate Colorectal Cancer Screening and Follow-up
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Kim, Dean at Penn State College of Medicine, Milton S. Hershey Medical Center
Other Study IDs: IRB19-1496; 1UG3CA233229 (NIH); 5UH3CA233229 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
Keywords: Multilevel intervention; Stepped wedge design; Implementation strategy; Federally qualified health center
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: The study participants included two federally qualified health centers (FQHCs) in Illinois and two in Indiana. Together, these four FQHCs had 65 primary care clinics and served 131,233 individual patients in 2020. One FQHC in Illinois and one FQHC in Indiana were randomly assigned to group 1, and the other two FQHCs were assigned to group 2. The only difference between the two groups was a 3-month delay in implementing the study intervention components.
  Interventions: Behavioral: Intervention Phase 1: Provider and Staff education; Behavioral: Intervention Phase 2: Provider and staff education + Patient reminder; Behavioral: Intervention Phase 3: Provider and Staff education + Patient reminder + Patient navigation
- Group 2: The study participants included two federally qualified health centers (FQHCs) in Illinois and two in Indiana. Together, these four FQHCs had 65 primary care clinics and served 131,233 individual patients in 2020. One FQHC in Illinois and one FQHC in Indiana were randomly assigned to group 1, and the other two FQHCs were assigned to group 2. The only difference between the two groups was a 3-month delay in implementing the study intervention components.
  Interventions: Behavioral: Intervention Phase 1: Provider and Staff education; Behavioral: Intervention Phase 2: Provider and staff education + Patient reminder; Behavioral: Intervention Phase 3: Provider and Staff education + Patient reminder + Patient navigation

INTERVENTIONS:
Behavioral: Intervention Phase 1: Provider and Staff education — In Phase 1, CRC control experts will identify critical messages on CRC, screening guidelines, and methods, and provide educational training to providers and staff in our partner FQHCs before implementing any intervention components. Additionally, the research team will provide refresher sessions and offer yearly training in CRC-relevant topics, including CRC and genetics.
Behavioral: Intervention Phase 2: Provider and staff education + Patient reminder — In Phase 2, we will add a patient reminder component using short message services (SMS) to engage and remind patients to complete the screening. For patients who use colonoscopy as a screening method, the SMS will also include instructions on bowel preparation and dietary restrictions for five days prior to the procedure.
Behavioral: Intervention Phase 3: Provider and Staff education + Patient reminder + Patient navigation — In Phase 3, we will add patient navigation services, which will address both organizational and individual barriers to obtaining screening.

SUMMARY:
Screening for colorectal cancer (CRC) not only detects disease early when treatment is more effective but also prevents cancer by finding and removing precancerous polyps. Because many of our nation's most disadvantaged and vulnerable individuals obtain health care at federally qualified health centers, these centers play a significant role in increasing CRC screenings among the most vulnerable populations. Furthermore, the full benefits of cancer screenings must include timely and appropriate follow-up of abnormal results. Thus, the purpose of this study is to implement a multilevel intervention to increase rates of CRC screenings, follow-ups, and referrals-to-care in federally qualified health centers (FQHCs). Also, we will examine the implementation strategies used to support the implementation process and their contribution to the adoption, implementation, and sustainment of the multilevel intervention. The multilevel intervention will target three different levels of influences: organization, provider, and individual. It will have multiple components, including provider and staff education, provider reminder, provider assessment and feedback, patient reminder, and patient navigation.

This study is a multilevel, three-phase, stepped wedge cluster randomized trial with four clusters of clinics from four different FQHCs. Our FQHC partners together have 40 primary care clinics and 130 primary care providers. During Phase 1, there will be a 3-month waiting period during which no intervention components will be implemented. After the 3-month waiting period, we will randomize two clusters of clinics to cross from the control to the intervention and the remaining two clusters to follow three months later. All clusters of clinics will stay at the same phase for nine months, followed by a 3-month transition period, and then cross over to the next phase. In Phase 1, we will implement provider and staff education sessions. In Phase 2, we will add provider reminders, patient reminders, and provider assessment and feedback. We will add patient navigation during the last phase.

Single level interventions are often insufficient at leading to sustainable changes. Multilevel interventions are needed to address multilevel contextual influences simultaneously. How to take advantage of multilevel interventions and how to implement such interventions and evaluate their effectiveness are the ultimate goals of this study.

DETAILED DESCRIPTION:
A. BACKGROUND

A1. Colorectal cancer control and FQHCs

Screening for CRC not only detects disease early when treatment is more effective but also prevents cancer by finding and removing precancerous polyps. Despite strong evidence to support CRC screening, nationally, only 68.8% of adults had up to date screening in 2018 [1]. This figure is even lower among racial/ethnic minorities and people who live in poverty [2-5]. Racial/ethnic minorities and people with low social-economic status often lack health insurance and a regular source of care. These populations also disproportionately receive health care in safety-net settings, such as federally qualified health centers (FQHCs) [6-7]. In 2018, FQHCs served 28 million patients, of whom 23% were uninsured, 63% were racial/ethnic minorities, and 91% were living below 200% poverty level [8]. Thus, FQHCs play a significant role in increasing CRC screening among the most vulnerable populations.

A2. Challenges of colorectal cancer control in FQHCs

Due to the cost and limited availability of specialty services combined with patient preferences, FQHCs often promote non-invasive screening methods, such as fecal occult blood test (FOBT) or fecal immunochemical tests (FIT), as the modality for screening [9-12]. To achieve the benefits of CRC screening using FOBT/FIT, timely follow-up of positive results must occur. While no national estimates of the proportion of individuals without follow-up diagnostic evaluation after receiving a positive FOBT/FIT exist, several studies report follow-up rates ranging from less than 50% to 90% within one year of a positive test [13-22], with integrated health care systems exhibiting higher follow-up rates by 12 months (82%-86%) compared to FQHCs (56%-58%) [23-24].

A3. Multilevel influences on cancer screening behavior

Individuals live and seek care in a complex environment, and multiple levels of contextual influences may affect individual decisions and actions [25-26]. Multilevel interventions target changes in more than one contextual level (e.g., organization, provider, and patient levels) to influence health behavior, health care practice, and health outcomes [27-28]. Although the call for multilevel interventions has increased [29-31], there is still a lack of evidence addressing how to implement multilevel interventions or how interventions at multiple levels interact and affect health outcomes.

B. STUDY OBJECTIVES

The overall objective of this study is to provide the evidence base for multilevel interventions that increase rates of CRC screening, follow-up, and referral-to-care at federally qualified health centers, and to understand how to improve the adoption, implementation, and sustainment of these interventions. In this study, we will test the effectiveness of our multilevel intervention while simultaneously observing and gathering information on the implementation process. The selection of our multilevel intervention components is based on extensive literature review, the strength of evidence, and findings from our previous studies and projects. The multilevel intervention will target three different levels of influence (organization, provider, and individual) to improve rates of CRC screening, follow-up, and referral-to-care at our partner FQHCs. Our multilevel intervention will have multiple components, including provider and staff education, provider reminder, provider assessment and feedback, patient reminder, and patient navigation.

The aims this study are fourfold: (1) use a stepped wedge design to implement a multilevel intervention in three phases, (2) collect quarterly data to track changes over time, (3) evaluate the implementation process and the effectiveness of implementation strategies through observations, interviews, and annual survey, and (4) evaluate the effectiveness of the multilevel intervention using multilevel and longitudinal modeling.

C. METHODS

CRC screening and follow-up processes are complex and include several steps and interfaces. However, very few interventional studies have simultaneously targeted patient-, provider-, and organization-level factors. Interventions that focus on reducing barriers across several levels will likely be more effective for increasing rates of CRC screening, follow-up, and referral-to-care.

C1. Multilevel Intervention and Implementation Strategy

Provider Level Component

Provider education

Numerous studies indicate the importance of physician recommendation in influencing a patient's CRC screening decision [31-44], and this factor is a primary predictor for patient adherence with screening guidelines [45-47]. The research team will provide tailored education and guidance on best practices for participating health professionals. The educational sessions will focus on CRC risk assessment, screening guidelines, cultural competency, shared decision making, and communication skills using an academic detailing approach. The academic detailing approach involves trained experts visiting health care professionals in their settings to provide tailored education and guidance on best practices, which have shown to have a significant effect on increasing rates of CRC screening [48-53]. Each session will last about 15 to 20 minutes and will take place during routine staff and provider meetings. These academic detailing sessions will be ongoing throughout the study period.

Provider assessment and feedback

We will combine academic detailing with practice facilitation, which includes assessment and feedback on aggregate and individual provider screening behavior and practice performance [54]. The reports will include CRC screening order rates, screening completion rates, follow-up rates for abnormal results, and referral to oncology care. Providers will be able to see each other's performances, which allows providers to compare and learn from each other's successes.

Provider reminder

Given the multitude of competing priorities during a patient encounter, CRC screening recommendations can be overlooked. A provider prompt generated electronically or manually by staff members will be implemented to remind providers to screen their eligible patients. Provider prompts have been shown to increase CRC screening rates [55].

C2. Organization and Individual Level Component

Patient reminder

Provider recommendation alone does not guarantee the completion of CRC screening, which involves patient compliance. We will implement a patient reminder component using a text-based platform, also known as short message service (SMS), to engage and remind patients to complete the screening. For patients who use colonoscopy as a screening method, the SMS will also include instruction on bowel preparation and dietary restrictions five days before the procedure. Studies have demonstrated that SMS patient reminders not only had a positive impact on screening rates but also improved the quality of bowel preparation [56-61].

Patient navigation

Patient navigation services will address both organization and individual influences. Patient navigation focuses on eliminating barriers by guiding a patient through a complex healthcare system, addressing education, sociocultural, and logistical needs using trained staff. We will hire and train two full-time CRC navigators and adapt and modify the well-studied New Hampshire Colorectal Cancer Screening Program (NHCRCSP) Patient Navigator Model [62-64].

C3. Implementation Strategy

The effectiveness of an intervention, in part, depends on the strength of the implementation process. We will conduct a pre-implementation organizational readiness assessment (ORA). We will use the Consolidated Framework for Implementation Research (CFIR) to guide our ORA. We will conduct key informant interviews with health system leadership and clinic leaders to evaluate: 1) current CRC screening workflow, 2) CRC data capturing and validation process, and 3) capacity and resources available to support the implementation. Also, we will conduct a readiness survey with clinical providers and support staff to assess organizational climate and culture. Our 29 survey items were adapted and modified from validated instruments65-68 that measured CFIR constructs using a Delphi method.

Effective strategies to support the implementation process is critical. Implementation strategies are actions taken to enhance the adoption, implementation, and sustainability of evidence-based interventions. We will use different implementation strategies to implement our multilevel intervention. Finally, we will implement our multilevel, multicomponent intervention in three phases along the CRC screening continuum. In Phase 1, we will collect baseline data and implement provider and staff education sessions. In Phase 2, we will add provider reminders, patient reminders, and provider assessment and feedback. We will add patient navigation during the last phase.

C4. Study Design

This study is a multilevel, three-phase, stepped wedge cluster randomized trial with four clusters of clinics from four different FQHCs. Our FQHC partners together have 40 primary care clinics and 130 primary care providers. During Phase 1, there will be a 3-month waiting period during which no intervention components will be implemented. After the 3-month waiting period, we will randomize two clusters of clinics to cross from the control to the intervention and the remaining two clusters to follow three months later. All clusters of clinics will stay at the same phase for nine months, followed by a 3-month transition period, and then cross over to the next phase. In Phase 1, we will implement provider and staff education sessions. In Phase 2, we will add provider reminders, patient reminders, and provider assessment and feedback. We will add patient navigation during the last phase.

C5. Study Sites

We will partner with four FQHCs, two in Illinois and two in Indiana. Together, our FQHC partners have 40 primary care clinics and 130 primary care providers and served 162,000 individual patients in 2018. Of the 162,000 patients, 78% were racial minorities, 93% live at or below 200% poverty, and 17% were uninsured. The CRC screening rates among our partners range from 25% to 43%.

C6. Process Evaluation

We will assess the potential causal and contextual factors that may be associated with observed outcomes at the provider and clinic levels. After completion of each phase, we will send all providers at our partner clinics a survey to assess their exposure to and experience with the intervention component. Furthermore, we will evaluate the changes in organizational culture and climate that may ascertain potential mechanisms of impact using the 29 survey items we developed based on the CFIR.

C7. Data Analysis Plan

We will conduct descriptive analyses, as well as within-group and between-group changes over time. Furthermore, to evaluate the four-component intervention effects, we will take a step-by-step approach. First, each intervention effect at each time phase will be estimated separately using linear-mixed effects models. The estimate of intervention effect in each model will be used to test if additional intervention component significantly affects outcome measures. Next, we will develop a grand model, including all intervention components simultaneously, in addition to the models described above.

ELIGIBILITY:
Eligibility for Federally Qualified Health Centers (FQHCs)

Inclusion criteria:

* Located in Illinois or Indiana
* Provide adult primary care
* Serve patients between the ages of 50 and 75 years
* Able to provide patient-level data

Exclusion criteria:

* Located outside Illinois or Indiana
* Do not provide adult primary care
* Unable to provide patient-level data

Eligibility for patients whom our FQHC partners serve:

Inclusion criteria:

* Between the ages of 50 and 75
* At general risk for colorectal cancer

Exclusion criteria:

* Patients who are younger than 45 years old or older than 75 years old
* Patients who are at high risk for colorectal cancer screening and require early screening before the age of 45

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are seen in our partner FQHCs, between the ages of 50 and 75 years old, and at general risk for colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kim, MD, Principal Investigator — University of Chicago
Locations (1):
- PCC Community Wellness Centers, Oak Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim K, Polite B, Hedeker D, Liebovitz D, Randal F, Jayaprakash M, Quinn M, Lee SM, Lam H. Implementing a multilevel intervention to accelerate colorectal cancer screening and follow-up in federally qualified health centers using a stepped wedge design: a study protocol. Implement Sci. 2020 Oct 29;15(1):96. doi: 10.1186/s13012-020-01045-4. PMID 33121536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited four federally qualified health centers (FQHCs): two in Illinois and two in Indiana. Together, these four FQHCs operate 65 primary care clinics and served 131,233 individual patients in 2020. One FQHC from each state was randomly assigned to Group 1, while the remaining two were assigned to Group 2. Both groups received the intervention; the only distinction was that implementation in Group 2 was delayed by three months compared to Group 1.
Units Other Than Participants: FQHCs
Groups:
- Group 1; Group 2: The study was conducted in four federally qualified health centers (FQHCs): two in Illinois and two in Indiana. One FQHC from Illinois and one from Indiana were randomly assigned to Group 1, and the remaining two formed Group 2. Both groups received all intervention components except that Group 2 began the intervention three months later than Group 1. The enrollment number reflects the total number of individual patients seen at each facility (FQHC) during each study phase. Because the study was conducted at the facility level, no individual consent or enrollment occurred. Additionally, the provider and staff education component was conducted at the facility (FQHC) level and did not target individual providers. Therefore, provider characteristics were not assessed at baseline and were not included in the Participant Flow or adverse event reporting.
  The intervention consists of three components:
  1. Provider and staff education,
  2. Patient reminders using short message services (SMS), and
  3. Remote patient navigation (PN).
  Implementation was phased as follows:
  * Phase 0: No intervention components, baseline data collection only
  * Phase 1: Component 1 only
  * Phase 2: Components 1 + 2
  * Phase 3: Components 1 + 2 +3
Period: Baseline (Months 0-12)
Arm/Group | Group 1 | Group 2
Started | 18099; 2 FQHCs | 20834; 2 FQHCs
Group 1 and Group 2 collect baseline data only, no intervention | 18099; 2 FQHCs | 20834; 2 FQHCs
Completed | 18099; 2 FQHCs | 20834; 2 FQHCs
Not Completed | 0; 0 FQHCs | 0; 0 FQHCs
Period: Step 1 (Months 13-18)
Arm/Group | Group 1 | Group 2
Started | 19318; 2 FQHCs | 18878; 2 FQHCs
Both Group 1 and Group 2 receive Component 1 (Provider and Staff Education) | 19318; 2 FQHCs | 18878; 2 FQHCs
Completed | 19318; 2 FQHCs | 18878; 2 FQHCs
Not Completed | 0; 0 FQHCs | 0; 0 FQHCs
Period: Step 2 (Months 19-21)
Arm/Group | Group 1 | Group 2
Started | 21102; 2 FQHCs | 15725; 2 FQHCs
Group 1 receives Component 2 (SMS Reminders) | 21102; 2 FQHCs | 0; 0 FQHCs
Completed | 21102; 2 FQHCs | 0; 0 FQHCs
Not Completed | 0; 0 FQHCs | 15725; 2 FQHCs
Not completed — In a 3-month delay period | 0 | 15725
Period: Step 3 (Months 22-30)
Arm/Group | Group 1 | Group 2
Started | 21102; 2 FQHCs | 15725; 2 FQHCs
Both Groups Receive Component 1 and Componet 2 | 21102; 2 FQHCs | 15725; 2 FQHCs
Completed | 21102; 2 FQHCs | 15725; 2 FQHCs
Not Completed | 0; 0 FQHCs | 0; 0 FQHCs
Period: Step 4 (Months 31-33)
Arm/Group | Group 1 | Group 2
Started | 21602; 2 FQHCs | 15037; 2 FQHCs
Group 1 receives all three components (provider and staff education+SMS Reminders+ Remote PN) | 21602; 2 FQHCs | 0; 0 FQHCs
Completed | 21602; 2 FQHCs | 0; 0 FQHCs
Not Completed | 0; 0 FQHCs | 15037; 2 FQHCs
Not completed — In a 3-month delay period | 0 | 15037
Period: Step 5 (Months 34-45)
Arm/Group | Group 1 | Group 2
Started | 21602; 2 FQHCs | 15037; 2 FQHCs
Both Groups Receive All Three Components | 21602; 2 FQHCs | 15037; 2 FQHCs
Completed | 21602; 2 FQHCs | 15037; 2 FQHCs
Not Completed | 0; 0 FQHCs | 0; 0 FQHCs

BASELINE CHARACTERISTICS:
Population: Patients who were between the ages of 50 and 75 at participating FQHCs during the Year 2020 (from January 1 to December 31), with FQHC 1 located in Illinois and FQHC 2 located in Indiana in each arm. The overall number of baseline participants was the total number of patients who were between the ages of 50 and 75 from both FQHC partners assigned to the Group.
Units Other Than Participants: FQHC
Groups:
- Group 1; Group 2: The study was conducted at 4 federally qualified health centers (FQHCs): 2 in Illinois and 2 in Indiana. One FQHC from Illinois and one from Indiana were randomly assigned to Group 1, and the remaining two formed Group 2. Both groups received all intervention components, except that Group 2 began the intervention 3 months later than Group 1. The enrollment number reflects the total number of individual patients seen at each facility (FQHC) during each study phase. Because the study was conducted at the facility level, no individual consent or enrollment occurred. Additionally, the provider and staff education component was conducted at the facility (FQHC) level. Therefore, provider characteristics were not assessed at baseline and were not included in the Participant Flow or adverse event reporting.
  The intervention consists of three components:
  1. Provider and staff education,
  2. Patient reminders using short message services (SMS), and
  3. Remote patient navigation (PN).
  Implementation was phased as follows:
  * Phase 0: No intervention components, baseline data collection only
  * Phase 1: Component 1 only
  * Phase 2: Components 1 + 2
  * Phase 3: Components 1 + 2 +3
  Baseline data collection was restricted to patients aged 50-75 years, the age group eligible for colorectal cancer screening in 2020. While provider and staff education sessions were part of the intervention components, no provider or staff characteristics were collected per protocol.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 18099 | 20834 | 38933
Number analyzed (FQHC) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Patients who were between the ages of 50 and 75 at each FQHC, with FQHC 1 in both groups located in Illinois and FQHC 2 in each group located in Indiana.
  years
    FQHC 1: number analyzed (Participants) | 8943 | 13906 | 22849
    FQHC 1 | 59.25 (6.272) | 58.77 (6.138) | 58.96 (6.195)
    FQHC 2: number analyzed (Participants) | 9156 | 6928 | 16084
    FQHC 2 | 60.04 (6.374) | 59.45 (6.126) | 59.79 (6.275)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Patients who were between the ages of 50 and 75 at each FQHC, with FQHC 1 in both groups located in Illinois and FQHC 2 in each group located in Indiana.
  Participants
    FQHC 1: number analyzed (Participants) | 8943 | 13906 | 22849
    FQHC 1: Male | 3338 | 5651 | 8989
    FQHC 1: Female | 5019 | 7478 | 12497
    FQHC 1: Unknown | 586 | 777 | 1363
    FQHC 2: number analyzed (Participants) | 9156 | 6928 | 16084
    FQHC 2: Male | 3806 | 2823 | 6629
    FQHC 2: Female | 5345 | 4105 | 9450
    FQHC 2: Unknown | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Patients who were between the ages of 50 and 75 at each FQHC, with FQHC 1 in both groups located in Illinois and FQHC 2 in each group located in Indiana.
  Participants
    FQHC 1: number analyzed (Participants) | 8943 | 13906 | 22849
    FQHC 1: Hispanic or Latino | 2811 | 3859 | 6670
    FQHC 1: Not Hispanic or Latino | 4882 | 8306 | 13188
    FQHC 1: Unknown or Not Reported | 1250 | 1741 | 2991
    FQHC 2: number analyzed (Participants) | 9156 | 6928 | 16084
    FQHC 2: Hispanic or Latino | 1295 | 664 | 1959
    FQHC 2: Not Hispanic or Latino | 4198 | 3316 | 7514
    FQHC 2: Unknown or Not Reported | 3663 | 2948 | 6611
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Patients who were between the ages of 50 and 75 at each FQHC, with FQHC 1 in both groups located in Illinois and FQHC 2 in each group located in Indiana.
  Participants
    FQHC 1: number analyzed (Participants) | 8943 | 13906 | 22849
    FQHC 1: American Indian or Alaska Native | 68 | 616 | 684
    FQHC 1: Asian | 75 | 177 | 252
    FQHC 1: Native Hawaiian or Other Pacific Islander | 34 | 75 | 109
    FQHC 1: Black or African American | 4440 | 5111 | 9551
    FQHC 1: White | 2332 | 4405 | 6737
    FQHC 1: More than one race | 716 | 1636 | 2352
    FQHC 1: Unknown or Not Reported | 1278 | 1886 | 3164
    FQHC 2: number analyzed (Participants) | 9156 | 6928 | 16084
    FQHC 2: American Indian or Alaska Native | 42 | 77 | 119
    FQHC 2: Asian | 66 | 93 | 159
    FQHC 2: Native Hawaiian or Other Pacific Islander | 11 | 28 | 39
    FQHC 2: Black or African American | 1317 | 1699 | 3016
    FQHC 2: White | 7217 | 4366 | 11583
    FQHC 2: More than one race | 193 | 66 | 259
    FQHC 2: Unknown or Not Reported | 310 | 599 | 909
Region of Enrollment [Number; unit: participants]
  United States | 18099 | 20834 | 38933
Colorectal Cancer (CRC) Screening Up-to-date Rate [Count of Participants; unit: Participants] — The number of patients between the ages of 50 and 75 who were up to date with CRC screening at each partner FQHC in 2020. Population: Number of patients who were between the ages of 50 and 75 and up to date with CRC screening at each FQHC in 2020.
  Participants
    FQHC 1: CRC Screening Up to Date: number analyzed (Participants) | 8943 | 13906 | 22849
    FQHC 1: CRC Screening Up to Date | 2998 | 2203 | 5201
    FQHC 2: CRC Screening Up to Date: number analyzed (Participants) | 9156 | 6928 | 16084
    FQHC 2: CRC Screening Up to Date | 4639 | 1817 | 6456
CRC Order Rate [Count of Participants; unit: Participants] — The number of patients between the ages of 50 and 75 who needed CRC screening and received a screening order at each partner FQHC. Population: Patients between the ages of 50 and 75 who needed an order for CRC screening at each FQHC in 2020.
  Participants
    FQHC 1: CRC Screening Order Rate: number analyzed (Participants) | 6493 | 12640 | 19133
    FQHC 1: CRC Screening Order Rate | 1804 | 3405 | 5209
    FQHC 2: CRC Screening Order Rate: number analyzed (Participants) | 5920 | 5399 | 11319
    FQHC 2: CRC Screening Order Rate | 3370 | 884 | 4254
CRC Screening Completion Rate [Count of Participants; unit: Participants] — The number of patients between the ages of 50 and 75 who needed CRC screening, received a screening order, and completed the screening at each partner FQHC in 2020. Population: Patients between the ages of 50 and 75 who needed CRC screening and received an order for screening at each FQHC in 2020.
  Participants
    FQHC 1: CRC Screening Completion Rate: number analyzed (Participants) | 1804 | 3405 | 5209
    FQHC 1: CRC Screening Completion Rate | 711 | 1320 | 2031
    FQHC 2: CRC Screening Completion Rate: number analyzed (Participants) | 3370 | 884 | 4254
    FQHC 2: CRC Screening Completion Rate | 1672 | 344 | 2016

OUTCOME MEASURES:

1. Primary Outcome: CRC Screening Rate
Description: The number of patients aged 50-75 years who were up-to-date with colorectal cancer screening during each implementation phase.
Time Frame: From date of randomization until the last subject completed the study. This could have been up to 36 months.
Population: The overall number represents all participants across all study phases. The number analyzed reflects only participants contributing data at the reported phase.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1; Group 2: The study was conducted in four federally qualified health centers (FQHCs): two in Illinois and two in Indiana. One FQHC from Illinois and one from Indiana were randomly assigned to Group 1, and the remaining two formed Group 2. Both groups received all intervention components except that Group 2 began the intervention three months later than Group 1.
  The intervention consists of three components:
  1. Provider and staff education,
  2. Patient reminders using short message services (SMS), and
  3. Remote patient navigation (PN).
  Implementation was phased as follows:
  * Phase 0: No intervention components
  * Phase 1: Component 1 only
  * Phase 2: Components 1 + 2
  * Phase 3: Components 1 + 2 +3
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 62022 | 49640
Participants
  Phase 1: Provider and Staff Education: number analyzed (Participants) | 19318 | 18878
  Phase 1: Provider and Staff Education | 8611 | 3989
  Phase 2: Provider Education + Patient Reminder: number analyzed (Participants) | 21102 | 15725
  Phase 2: Provider Education + Patient Reminder | 9438 | 3186
  Phase 3: Provider and Staff Education + Patient Reminders + Remote Patient Navigation: number analyzed (Participants) | 21602 | 15037
  Phase 3: Provider and Staff Education + Patient Reminders + Remote Patient Navigation | 10720 | 3303

2. Primary Outcome: CRC Screening Ordering Rate
Description: The number of patients between the ages of 50 and 75 who needed CRC screening and received a screening order (excluding participants who received an order but have already been up to date with screening ) during each implementation phase.
Time Frame: From date of randomization until the date subject completed the study. This could have been up to 36 months.
Population: The overall number represents all participants who needed screening across all study Phases. The number analyzed reflects only participants contributing data at the reported phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 41263 | 43243
Participants
  Phase 1: Provide and Staff Education: number analyzed (Participants) | 13403 | 16451
  Phase 1: Provide and Staff Education | 7012 | 5087
  Phase 2: Provider and Staff Education + Patient Reminders: number analyzed (Participants) | 14180 | 13769
  Phase 2: Provider and Staff Education + Patient Reminders | 6458 | 4757
  Phase 3: Provide and Staff Education + Patient Reminders + Remote Patient Navigation: number analyzed (Participants) | 13680 | 13023
  Phase 3: Provide and Staff Education + Patient Reminders + Remote Patient Navigation | 6478 | 4611

3. Primary Outcome: CRC Screening Completion Rate
Description: The number of patients between the ages of 50 and 75 who needed CRC screening, received an order for screening, and completed the screening during each implementation phase.
Time Frame: From date of randomization until the date subject completed the study. This could have been up to 36 months.
Population: The overall number represents all participants who needed CRC screening and received an order across all study phases. The number analyzed reflects only participants contributing data at the reported milestone.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 19948 | 14455
Participants
  Phase 1: Provider and Staff Educatioin: number analyzed (Participants) | 7012 | 5087
  Phase 1: Provider and Staff Educatioin | 3106 | 1917
  Phase 2: Provider and Staff Education + Patient Reminders: number analyzed (Participants) | 6458 | 4757
  Phase 2: Provider and Staff Education + Patient Reminders | 3031 | 1749
  Phase 3: Provider and Staff Education + Patient Reminders + Remote Patient Navigation: number analyzed (Participants) | 6478 | 4611
  Phase 3: Provider and Staff Education + Patient Reminders + Remote Patient Navigation | 3278 | 1691

4. Secondary Outcome: Provider Education Participation
Description: The number of providers who attended the annual education sessions during Phase 1 and Phase 2. To accommodate the COVID-19 restrictions, all sessions were delivered via Zoom, with multiple sessions scheduled within each FQHC based on clinic availability. Both groups received the education component simultaneously, with no delay in implementation.
Time Frame: From the date of the first education session until the completion of the last education sessions. This could have been up to 24 months.
Population: The overall number represents the total number of providers invited to the education sessions during Phase 1 and Phase 2. The number analyzed reflects the number of providers invited to the education sessions during the reported phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 527 | 340
Participants
  Phase 1: Provider and Staff Education: number analyzed (Participants) | 255 | 176
  Phase 1: Provider and Staff Education | 129 | 44
  Phase 2: Provider and Staff Education + Patient Reminders: number analyzed (Participants) | 272 | 164
  Phase 2: Provider and Staff Education + Patient Reminders | 126 | 89

5. Secondary Outcome: Patient Reminder Enrollment
Description: The number of participants who received a FIT or colonoscopy order (excluding Cologuard, which provides its own reminder services) and subsequently enrolled in the short message service (SMS) reminder system during Phase 2 and Phase 3. The SMS platform was used to engage participants and remind them to complete their screenings; participants could opt out at any time by replying "STOP".
Time Frame: From the initiation of the SMS reminder system until the last participant enrolled. This could have been up to 30 months.
Population: The overall number represents the total number of participants who received a FIT or colonoscope order during the implementation of Phase 1 and Phase 2. The number analyzed reflects only the number of participants contributing data to the reported milestone.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 13013 | 10824
Participants
  Phase 2: Provider and Staff Education + Patient Reminders: number analyzed (Participants) | 6628 | 5464
  Phase 2: Provider and Staff Education + Patient Reminders | 4756 | 4693
  Phase 3: Provider and Staff Education + Patient Reminders + Remote Patient Navigation: number analyzed (Participants) | 6385 | 5360
  Phase 3: Provider and Staff Education + Patient Reminders + Remote Patient Navigation | 5198 | 3943

6. Secondary Outcome: Impact of Remote Patient Navigation Services
Description: The number of participants who received remote navigation services (phone-based navigation) during Phase 3 and subsequently completed their screenings.
Time Frame: From the navigation service initiated at the partner FQHC until the completion of the study, assessed up to 16 months.
Population: The overall number represents the number of participants whom the navigators successfully contacted and spoke to during Phase 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 1330 | 1127
Participants | 529 | 284

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from the beginning of the study, following the recruitment of the first participating federally qualified health center in 2020, and continued until December 2023, when the study was completed. Up to a total of four years of adverse events were monitored, and adverse event data were collected from each FQHC during each of the implementation phases.
Description: We followed the definitions as described by clinicaltrials.gov to monitor adverse events and collect relevant data at each FQHC.
Groups:
- Group 1 During Phase 0 (No Intervention); Group 2 During Phase 0 (No Intervention): The study was conducted in four federally qualified health centers (FQHCs): two in Illinois and two in Indiana. One FQHC from Illinois and one from Indiana were randomly assigned to Group 1, and the remaining two formed Group 2. Both groups received all intervention components except that Group 2 began the intervention three months later than Group 1. The enrollment number reflects the total number of individual patients seen at each facility (FQHC) during each study phase. Because the study was conducted at the facility level, no individual consent or enrollment occurred. Additionally, the provider and staff education component was conducted at the facility (FQHC) level and did not target individual providers. Therefore, provider characteristics were not assessed at baseline and were not included in the Participant Flow or adverse event reporting.
  The intervention consists of three components:
  1. Provider and staff education,
  2. Patient reminders using short message services (SMS), and
  3. Remote patient navigation (PN).
  Implementation was phased as follows:
  * Phase 0: No intervention components
  * Phase 1: Component 1 only
  * Phase 2: Components 1 + 2
  * Phase 3: Components 1 + 2 +3
- Groups 1 During Phase 1; Groups 2 During Phase 1: In Phase 1, only Component 1 (provider and staff education) was implemented.
- Group 1 During Phase 2; Group 2 During Phase 2: In Phase 2, Component 2 (patient reminders) was added in addition to Component 1.
- Group 1 During Phase 3; Group 2 During Phase 3: In Phase 3, all three intervention components (provider and staff education + patient reminders + remote patient navigation) were implemented.
Arm/Group | Group 1 During Phase 0 (No Intervention) | Group 2 During Phase 0 (No Intervention) | Groups 1 During Phase 1 | Groups 2 During Phase 1 | Group 1 During Phase 2 | Group 2 During Phase 2 | Group 1 During Phase 3 | Group 2 During Phase 3
All-Cause Mortality (participants affected / at risk) | 0/18099 | 0/20834 | 0/19318 | 0/18878 | 0/21102 | 0/15725 | 0/21602 | 0/15037
Serious Adverse Events (participants affected / at risk) | 0/18099 | 0/20834 | 0/19318 | 0/18878 | 0/21102 | 0/15725 | 0/21602 | 0/15037
Other Adverse Events (participants affected / at risk) | 0/18099 | 0/20834 | 0/19318 | 0/18878 | 0/21102 | 0/15725 | 0/21602 | 0/15037

LIMITATIONS AND CAVEATS:
Relevant colorectal screening data, including up-to-date screening rates, screening order rates, and completion rates, were extracted from the electronic health records. However, each participating federally qualified health center used a different EMR system, and the capability to extract relevant data was sometimes limited by the system in use, particularly in one of the participating FQHCs, which used an older system and was unable to extract some data elements successfully.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT04514341/Prot_SAP_000.pdf